CLINICAL TRIAL: NCT04100642
Title: A Phase I Clinical Study Assessed the Safety Tolerance and Pharmacokinetic Characteristics of Hemay808 in Healthy Adult Volunteers
Brief Title: A Phase I Clinical Study of Hemay808
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YQ-M-18-08
Record Dates: First submitted 2019-05-20; First posted 2019-09-24 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2019-09

CONDITIONS: Safety Issues
Keywords: first in human; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1% Hemay808 apply to 25%BSA (Active Comparator): 8 subjects use 1% Hemay808
  Interventions: Drug: Hemay808
- 3% Hemay808 apply to 25%BSA (Experimental): 8 subjects use 3% Hemay808
  Interventions: Drug: Hemay808
- 3% Hemay808 apply to 55%BSA (Experimental): 6 subjects use 3% Hemay808
  Interventions: Drug: Hemay808
- 7% Hemay808 apply to 25%BSA (Experimental): 8 subjects use 7% Hemay808
  Interventions: Drug: Hemay808
- placebo apply to 25%BSA (Placebo Comparator): 6 subjects use placebo apply to 25%BSA
  Interventions: Drug: Placebo
- placebo apply to 55%BSA (Placebo Comparator): 2 subjects use placebo apply to 55%BSA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemay808 — topical apply
  Arms: 1% Hemay808 apply to 25%BSA; 3% Hemay808 apply to 25%BSA; 3% Hemay808 apply to 55%BSA; 7% Hemay808 apply to 25%BSA
Drug: Placebo — topical apply
  Arms: placebo apply to 25%BSA; placebo apply to 55%BSA

SUMMARY:
This is a first-in-human study in health volunteers. The purpose is the local tolerability and systemic safety of Hemay808, which is an ointment made of a novel small molecule Hemay028. The safety and systemic pharmacokinetics (PK) of Hemay028 will be evaluated following topical application of Hemay808 to healthy volunteers.

DETAILED DESCRIPTION:
There are two pre-test groups. Group1 use Hemay808 and placebo on sensitive areas. Group2 will only topical use Hemay808 on 5%BSA.

After 2 pre-test group, 4 formal testing groups will start. 1% Hemay808 apply to 25%BSA; 3% Hemay808 apply to 25%BSA; 3% Hemay808 apply to 55%BSA; 7% Hemay808 apply to 25%BSA. First a single doses then wash-out for three days, after that subjects will applicant twice daily for 7 days to assess the local skin tolerability, and systemic PK of these treatments.

Approximately 42 healthy adult volunteers will be enrolled in this study with 8- 10 volunteers each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects aged ≥ 18 to 45 years, inclusive.
* Male weight 50kg during screening; Female weight 45kg; Body mass index (BMI) between 19 and 24kg/m2 (including boundary value).
* No ulceration, injury, sunburn, redness, rash, pigmentation, uneven skin color, excessive freckles or abnormal fever were found in the skin of the target coating area during screening and before administration.
* Chinese health volunteers
* Women of child-bearing age and all male subjects must undertake to take effective contraceptive measures during the study period and within 6 months after discontinuation of the medication.
* All subjects will voluntarily participate in the study after knowing the content of the study and possible adverse drug reactions (ADR), and must sign the informed consent approved by the ethics committee before starting to accept any inspection specified in this study.
* Subjects will be able to communicate well with the investigator and promise to complete the study in accordance with the study regulations.

Exclusion Criteria:

* History of mental illness or a genetic history of mental illness, or a history of serious (5.0 NCI CTCAE 3) cardiovascular, liver, kidney, digestive tract, neurological or other diseases.
* Any dermatological condition other than atopic dermatitis that in the Investigator's opinion may interfere with the evaluation of the patient's atopic dermatitis.
* History of atopic dermatitis.
* History of severe (5.0 NCI CTCAE 3) skin disease.
* Current diagnosis or history allergic disease (such as allergic nose pharynx, allergic asthma), has a history of drug allergy, always have a skin allergy (including but not limited to allergic to the patch, for metal, cosmetics and household items with contact dermatitis), known to gao min physique, or known or the judge may, the active ingredient to the study drug has allergies or accessories.
* Regular smoking (>5 / day) or drinking (>28 units/day); Unit: 285mL beer or 25mL spirits or 100mL wine); Or drink too much tea every day (>15g tea/day); Generally, each time tea is brewed (3~5g of tea), coffee or drinks containing caffeine (>500mg/ day) (one cup of coffee contains about 85mg of caffeine).
* Subjects were not negative by virological examination (hepatitis b surface antigen, hepatitis c antibody, human immunodeficiency virus) and gelagglutination test of treponema pallidum.
* Common drugs (MDMA, MOR, MAMP, KETA) did not meet the requirements.
* Have major surgery within 2 months prior to screening, or have any surgery within 4 weeks prior to screening.
* Had treated cancer within 5 years prior to screening (except for squamous cell, basal cell, or in situ skin cancers that were cured only by cryopreservation or surgical excision).
* History of use (including topical use) for any reason within 2 weeks prior to administration. Except the investigator determines that the drug used has a half-life of >5 years after the start of this study, the corresponding subjects can also be enrolled.
* Have a history of drug abuse or drug abuse, or regularly (>3 times/week within 3 months before screening) use Chinese herbs, tranquilizers, sleeping pills, tranquilizers and other addictive drugs.
* Participated in any clinical trial within 3 months prior to screening.
* Non-physiologic blood loss 400ml (including trauma, blood collection and blood donation) within 3 months prior to screening, or blood donation during the study period or within 1 month after the study.
* The female subjects were in lactation or pregnancy at the time of screening (meaning the serum human chorionic gonadotropin test results of female subjects of child-bearing age were higher than the reference value).
* Female subjects with menstrual disorders for the last 2 months.
* Female subjects of reproductive age had unprotected sex with a heterosexual partner within 14 days prior to screening.
* Subjects of child-bearing age (male or female) plan to become pregnant during or within 6 months after the end of the study.
* Other circumstances in which the researcher considers it inappropriate to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events. | Day 1 to Day 30
  Incidence of AEs

SECONDARY OUTCOMES:
Cmax | pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 14, 24, 36, 48, 72 hours post-dose
  Maximum observed plasma concentration.
Tmax | pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 14, 24, 36, 48, 72 hours post-dose
  Time of maximum concentration Time of maximum concentration Time of maximum concentration Time of maximum concentration Time of maximum concentration Time of maximum concentration Time of Time of maximum concentration Time of maximim plasma concentration
AUCt | pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 14, 24, 36, 48, 72 hours post-dose
  Area under the plasma concentration-time curve from time zero extrapolated to infinity.
AUC∞ | pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 14, 24, 36, 48, 72 hours post-dose
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermotology hospital, Chinese academy of medical science, Nanjing, Jiangsu, China